CLINICAL TRIAL: NCT04940936
Title: Shared Decision Making on Radiation Dose for Stereotactic Body Radiotherapy of Malignancies Located Less Than 1 cm From the Thoracic Wall. A Randomized Trial
Brief Title: Shared Decision Making on Radiation Dose for Lung Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SDM Lung SBRT
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Decision Making, Shared; Stereotactic Body Radiation Therapy; Lung Cancer, Non-small Cell; Radiation Toxicity; Lung Metastases
Keywords: Stereotactic body radiation therapy; Lung malignancy; Shared decision making; Patient Decision Aid
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: After inclusion in the study, the patients are randomized into Arm A and B as follows:
  Arm A: Consultation as usual. Patients are informed about treatment and the two dose options according to current standards and routines.
  Arm B: Consultation using the PtDA. Patients are informed about treatment and dose options using the PtDA to make the pros and cons clearer to the patients.
  The doctors and nurses in the Radiotherapy Department will be educated in the use of the PtDA before initiation of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - control (No Intervention): The patients are offered high or lower dose according to usual practice
- B - Intervention (Experimental): The Patient Decision Aid is used during the consultation to aid in the decision on high or lower dose.
  Interventions: Behavioral: A Patient Decision Aid

INTERVENTIONS:
Behavioral: A Patient Decision Aid — The Patient Decision Aid informs about the pros and cons of each option
  Arms: B - Intervention

SUMMARY:
A Patient Decision Aid (PtDA) is developed during a workshop in close collaboration with selected patients. The PtDA is subsequently used in the consultation between patient and physician to facilitate their shared decision on the dose of stereotactic body radiation therapy (SBRT) for lung tumors located less than 1 cm from the thoracic wall.

Hypothesis: The use of a PtDA will increase the extent of Shared Decision Making (SDM) during the consultation and result in patients being more directly involved in the planning of their treatment.

DETAILED DESCRIPTION:
When a lung tumor is located close to the thoracic wall, there is an increased risk of developing chest wall pain or rib fracture following SBRT of the tumor. A meta-analysis has shown the pooled risk of chest wall pain to be 11% and that of rib fracture to be 6.3% with significant differences between individual studies. These side effects may occur several years after the treatment.

SDM is a collaborative process allowing patients and healthcare professionals to make decisions together taking into account the best scientific evidence as well as patients' values, preferences, life situation, and knowledge about disease process and prognosis.

PtDAs are tools designed to assist caregivers in the process of informing patients about relevant treatment options. PtDAs contain factual and balanced information about the options and the pertaining pros, cons, and probabilities. The tools are relevant when the decision is preference-sensitive, that is, the right treatment cannot be decided based on professional knowledge alone. The use of PtDAs has shown to provide a number of positive effects on the patients, including increased knowledge of options, better understanding of risks, and clarity as to what matters most in their life situation. Other effects are decreased decisional conflict and a higher degree of involvement in decision making.

This is a randomized trial enrolling eligible patients during a period of 16 months. SDM will be used in the planning of SBRT to patients with peripheral non-small cell lung tumors or lung metastases and offer them the choice between high (66 Gy in 3 fractions) and low (45 Gy in 3 fractions) radiation dose.

A total of 40 patients will be included in the study, i.e. 20 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed or high probability of non-small cell lung cancer, or metastasis from other cancer, located ≤ 1 cm from the thoracic wall. High probability refers to consensus on the diagnosis at the local multi-disciplinary lung tumor conference.
* Eligible for stereotactic body radiation therapy in ablative doses (i.e. 66/45 Gy in 3 fractions) following national guidelines (2).
* Can read and understand Danish.
* Written and orally informed consent.
* Performance status 0-2
* Life expectancy > 6 months assessed by the physician during the consultation.

Exclusion Criteria:

* Previous radiation therapy in the thoracic region (lung, breast or mediastinum), if it is not possible to produce a new radiation plan of 66 or 45 Gy in 3 fractions that considers previous radiation therapy and still complies with all constraints, including dose to the thoracic wall. Previous surgery in the thorax is allowed.
* Mental or social conditions preventing full understanding of the information or the planned treatment and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
The extent of shared decision making in the consultation between patient and oncologist as measured by the OPTION tool | During the one hour primary consultation.
  Minimum value: 0. Maximum value: 48. The higher the value, the higher the extent of SDM during the consultation

SECONDARY OUTCOMES:
Difference in patient perceived level of shared decision making between arm A and B as measured by the tool SDM-Q9. | Immediately after the primary consultation
  Minimum value 0. Maximum value 45. The higher the value, the higher the patient experienced extent of SDM during the consultation
Difference in patient perceived level of shared decision making between arm A and B as measured by the tool SDM_P4 | Immediately after the primary consultation
  Minimum value 0. Maximum value 4. The higher the value, the higher the patient experienced extent of SDM during the consultation
Difference in patient perceived level of shared decision making between arm A and B as measured by the tool CollaboRATE | Immediately after the primary consultation
  Minimum value 0. Maximum value 27. The higher the value, the higher the patient experienced extent of SDM during the consultation
Difference in decisional conflict between patients in arm A and B as measured by the Decision Conflict Scale | Immediately after the primary consultation
  Minimum value: 0. Maximum value: 64. The higher the value, the more decisional conflict.
Difference in decisional regret between patients in arm A and B as measured by the Decision Regret Scale | Reported by the patients six months and 3 years after the primary consultation
  Minimum value: 5. Maximum value: 25. The higher the value, the more decisional regret.
Difference in fear of cancer recurrence between patients in arm A and B as measured by the Fear of Cancer Recurrence - Short Form questionnaire | Reported by the patients six months and 3 years after the primary consultation
  Minimum value: 0. Maximum value: 36. The higher the value, the more fear of recurrence.
Number of patients developing chest wall pain and/or rib fracture during the 5-year follow-up program | Up to 5 years
  Evaluated by the physician every three months the first two years and then every six months the following three years.
Quality of Life as measured by the questionnaire EORTC QLQ-C30. | Up to 5 years
  Thirty questions with two different scales (1-4 and 1-7). The higher the value, the more symptoms/problems.
  Completed by the patients every three months the first two years and then every six months the following three years.
Quality of Life as measured by the questionnaire EORTC QLQ-LC29 | Up to 5 years
  Twenty-nine questions on a scale from 1 to 4. The higher the value, the more symptoms/problems.
  Completed by the patients every three months the first two years and then every six months the following three years.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Fink, MD, Principal Investigator — Department of Oncology, Vejle Hospital
Locations (1):
- Vejle Hospital, Department of Oncology, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be available on relevant request.

REFERENCES:
- [Derived] Fink TL, Hansen TF, Kristiansen C, Hansen TS, Thing RS, Timm S, Steffensen KD. Enhancing patient engagement: the influence of an in-consult patient decision aid on shared decision-making for lung tumour radiation - protocol for the randomised trial 'SDM Lung SBRT'. BMJ Open. 2025 Jan 20;15(1):e088595. doi: 10.1136/bmjopen-2024-088595. PMID 39833001